CLINICAL TRIAL: NCT00697437
Title: Effect of Ketoconazole Inhibition of CYP3A on Urinary Excretion of Docetaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr Goh Boon Cher, National University Hospital, Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK01/01/06
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Docetaxel; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- docetaxel only (Experimental)
  Interventions: Drug: Docetaxel
- docetaxel with ketoconazole (Experimental)
  Interventions: Drug: Docetaxel; Drug: Ketoconazole

INTERVENTIONS:
Drug: Docetaxel — 70mg q3wx 1 dose
Drug: Ketoconazole — 6 doses of oral ketoconazole 200mg bid starting 2 days before, and with 1 dose to be completed after, docetaxel infusion
  Arms: docetaxel with ketoconazole

SUMMARY:
Primary Objective:

* To confirm if ketoconazole inhibition of CYP3A activity affects fractional excretion of docetaxel in the urine.

Secondary Objective:

* To compare the metabolite ratios of the major metabolites of docetaxel in the presence and absence of CYP3A inhibition.

DETAILED DESCRIPTION:
Introduction: This is a follow-up protocol to an earlier study entitled "A phase I study of docetaxel with ketoconazole modulation in solid tumors" (PH14/01) which showed 2-fold reduction in docetaxel clearance and a clear correlation with renal function.

Aims: The aim of this study is to confirm that ketoconazole inhibition of CYP3A activity changes the urinary excretion profile of docetaxel.

Methodology: This is a single-centre, crossover study. Ten patients (calculated sample size =5, α=0.05, β=0.8, difference in means=5%, within group standard deviation=3) will be accrued and randomly assigned to receive docetaxel at either 75mg/m2 q3w x 1 dose or 70mg q3w x 1 dose with ketoconazole 200mg bid x q3d at cycle 1 of chemotherapy. This will be followed by a 20-day washout period before receiving the other regimen of docetaxel at cycle 2. Blood samples of 5mls each will be drawn at times 0, 0.5h, 1h, 1.5h, 3h, 4h, 6h and 24h after the onset of docetaxel infusion for pharmacokinetics analysis. A 24-hour urine collection commencing on the same day as docetaxel infusion will be required of the patients. All urine over the next 24 hours must be collected and returned to the study coordinator on Day 2 of each study cycle for docetaxel analysis and creatinine clearance determination. The amount of docetaxel excreted by each patient with and without ketoconazole modulation will be determined by a LCMSMS method and compared.

Clinical Relevance: This is to ensure the safe advocation of a dose-sparing strategy established in an earlier study for the costly agent docetaxel by confirming if changes in excretion profile occurs once its major route of hepatic metabolism is blocked.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which docetaxel is indicated.
2. Patients must have measurable or evaluable disease.
3. With the exception of alopecia, fatigue, nausea and asthenia, patients must have resolution of all acute toxic effects of any prior surgery' radiotherapy or chemotherapy to National Cancer Institute (NCI) Common Toxicity Criteria version 3.0 grade < 1.
4. Patients must have ECOG performance status ≤ 2 (Karnofsky ≥ 60%).
5. Patients must have a life expectancy of greater than 3 months.
6. Patients must have normal renal and marrow function as defined below:

   * leukocytes ≥ 3,000/μl
   * absolute neutrophil count ≥ 1,500/μl
   * platelets ≥ 100,000/μl
   * haemoglobin ≥ 7g/dL
   * creatinine ≤ 1.5 X institutional upper limit of normal
7. Patients with abnormal liver function tests (AST/ALT ≤ 3 x institutional upper limits of normal; ALP ≤ 5x ULN; total bilirubin ≤ 2x ULN) will be eligible for enrollment.
8. Patients must have adequate renal functions (serum creatinine within normal laboratory limits).
9. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents.
3. Patients who have rapidly progressive intracranial or spinal metastatic disease (including patients who require corticosteroid for CNS disease).
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or ketoconazole used in study.
5. Patients who have prior medications known to be metabolized by or induce/inhibit CYP3A4 within 1 week of each treatment cycle.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because docetaxel is embryotoxic/fetotoxic with the potential for abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with docetaxel, breastfeeding should be discontinued if the mother is treated with docetaxel. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To confirm if ketoconazole inhibition of CYP3A activity affects fractional excretion of docetaxel in the urine. | 9 weeks

SECONDARY OUTCOMES:
To compare the metabolite ratios of the major metabolites of docetaxel in the presence and absence of CYP3A inhibition. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Goh BC, Lee SC, Wang LZ, Fan L, Guo JY, Lamba J, Schuetz E, Lim R, Lim HL, Ong AB, Lee HS. Explaining interindividual variability of docetaxel pharmacokinetics and pharmacodynamics in Asians through phenotyping and genotyping strategies. J Clin Oncol. 2002 Sep 1;20(17):3683-90. doi: 10.1200/JCO.2002.01.025. PMID 12202670
- [Background] Tham LS, Goh BC, Wang LZ, Yong WP, Wong CI, Lee SC, Soo R, Sukri N, Lee HS. Ketoconazole inhibition of CYP3A activity made midazolam but not docetaxel pharmacokinetics more predictable. (Abstr) 2006 American Society for Clinical Pharmacology and Therapeutics Annual Meeting (Baltimore, MD).